CLINICAL TRIAL: NCT04037111
Title: Clinical Study of Escitalopram Oxalate Combined With Transcutaneous Vagus Nerve Stimulation in the Treatment of Depression and Concomitant Inflammatory Symptoms
Brief Title: Clinical Study of Escitalopram Oxalate Combined With taVNS in Depression and Concomitant Inflammatory Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 82554333
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Major Depressive Disorder; Rheumatoid Arthritis
MeSH Terms: conditions — Depressive Disorder, Major; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- drug treatment and active VNS (Experimental): At the same time, actice VNS, escitalopram oxalate tablets were treated for 2 months.
  Interventions: Device: Transcutaneous electrical vagus nerve stimulation; Drug: drug treatment
- drug treatment and sham VNS (Sham Comparator): It received oxacillin oxalate tablets and sham VNS for 2 months.
  Interventions: Device: Sham vagus nerve stimulation; Drug: drug treatment
- drug treatment (Other): The dose of escitalopram oxalate tablets was maintained at 10-20mg/ day without VNS stimulation.
  Interventions: Drug: drug treatment

INTERVENTIONS:
Device: Transcutaneous electrical vagus nerve stimulation — The patient received active VNS and escitalopram oxalate tablets for 2 months.When the VNS was stimulated, the two electrodes were vertically attached to the left carotid sinus at 2cm, or the auricular clip electrode was applied to the tragus.
  Other Names: VNS stimulated once a day for 30 minutes each time with a stimulating intensity of 1-2 mA.
  Arms: drug treatment and active VNS
Device: Sham vagus nerve stimulation — The patient received sham VNS.When the VNS was stimulated, the two electrodes were vertically attached to the left carotid sinus at 2cm, or the auricular clip electrode was applied to the tragus.
  Arms: drug treatment and sham VNS
Drug: drug treatment — Escitalopram oxalate tablets should be taken orally once every morning for 2 months, each time 10-20mg

SUMMARY:
This study is expected to include 90 patients with major depressive disorder and rheumatoid arthritis as study subjects.Randomly divided into 3 groups: drug + VNS stimulation group, drug + sham stimulation group and drug group, each group had 30 patients.The treatment period of each group was 8 weeks.Age and sex were matched in all three groups.Scale evaluation and inflammatory factor test were performed before treatment (baseline), at week 4 and week 8 after treatment.Head MRI, evoked potential, and electrocardiogram were performed at baseline and at the end of week 8.

DETAILED DESCRIPTION:
1. Drug +VNS stimulation group: both VNS and escitalopram oxalate tablets were treated for 2 months. VNS stimulation was treated once a day for 30 minutes at the intensity of 1-2mA. Drug treatment: the dose of escitalopram oxalate tablets was maintained at 10-20 mg/ day
2. Drug + sham stimulation group: the patients were treated with escitalopram oxalate tablets and sham VNS for 2 months. Sham VNS stimulation: the sham stimulation device automatically stops after 30 seconds of stimulation. Drug treatment was the same as the above group.
3. Drug group: the dose of escitalopram oxalate tablets was maintained at 10-20 mg/ day without VNS stimulation

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old, in accordance with DSM-5 diagnostic criteria for major depressive disorder, or meet the diagnostic criteria for rheumatoid arthritis. The major depressive disorder is first or at least not used in the 5 half-life of the drug. Antidepressants, antipsychotics or anticonvulsants.
* Hamilton Depression Rating Scale (HAMD) 17 scores over 17 points.

Exclusion Criteria:

* Brain organic lesions (such as cerebral hemorrhage, large area cerebral infarction, encephalitis, epilepsy); cardiac QTc interval > 450ms;
* Currently or have been diagnosed with other major diseases (such as coronary heart disease, pulmonary heart disease, etc.)
* Those who are currently or have been diagnosed with other mental disorders other than major depressive disorder (except for anxiety disorder);
* Patients who have a serious risk of suicide or who have had suicide attempts;
* Those who are using or have been treated with escitalopram oxalate are not effective;
* Those who are participating in or have participated in vagus nerve or transcranial electrical stimulation for less than 3 months;
* MRI scan taboos and high-risk groups;
* Pregnancy, breastfeeding or planning for pregnancy during the trial;
* Refusal to sign informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Changes of Hamd-17 Scale Scores From Baseline to Week 8 | From the baseline to the week 8
  After 8 weeks of treatment, the rate of hamd-17 scale score was decreased compared with the baseline

SECONDARY OUTCOMES:
Changes of Hamd-17 Scale Scores from Baseline to Week 4 | From baseline to week 4
  Changes of hamd-17 scale scores from baseline to the end of treatment at week 4
Changes of MADRS Scale and SDS Scale Score from Baseline to Week 4 and Week 8 | From baseline to week 4 and week 8
  Changes of MADRS SDS scale scores from baseline after the end of treatment at week 4 and week 8
The Clinical Improvement Rate at Week 4 and Week 8 | From baseline to week 4 and week 8
  Clinical improvement rates at week 4 and 8 (50% reduction in hamd-17 or MADRS from baseline)
The Remission Rate after 8 Weeks' Treatment | From baseline to week 8
  Hamd-17 or MADRS scores are less than or equal to 7
Changes of Cytokines from Baseline to Week 4 and Week 8 | From baseline to week 4 and week 8
  Changes in cytokines such as TNF-α, IL-γ, IL-4, IL-8 and IL-10 from baseline to the end of treatment after week 4 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Jin Sun, Principal Investigator — Xidian University, School of Life Science and Technology
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No